CLINICAL TRIAL: NCT06529497
Title: Efficacy of Racecadotril in Addition to Standard Treatment i in Decreasing the Duration of Acute Diarrhoea in Children as Compared to Standard of Treatment Alone
Brief Title: Racecadotril Versus Standard Treatment in Decreasing the Duration of Acute Diarrhoea in Children
Acronym: ERADICATE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Aqsa Jabeen, Consultant, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-30/RMU
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Diarrhoea
Keywords: Stool; Diarrhoea; Paediatrics
MeSH Terms: conditions — Diarrhea | interventions — racecadotril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group receiving (racecadotril+ORS+Zinc) (Experimental): The intervention group will receive racecadotril+ORS+Zinc while the reference group will receive ORS+Zinc alone
  Interventions: Drug: Racecadotril
- the control group (receiving ORS + Zinc or standard treatment) (Active Comparator): The intervention group will receive racecadotril+ORS+Zinc while the reference group will receive ORS+Zinc alone
  Interventions: Drug: Racecadotril

INTERVENTIONS:
Drug: Racecadotril — The intervention group will receive racecadotril+ORS+Zinc
  Other Names: ORS+Zinc

SUMMARY:
Acute watery diarrhea is defined as the passage of 3 or more loose or liquid stools per day for 3 or more days but less than 14 days, including patients with mild to moderate dehydration per WHO classification. The study's outcome variables are stool frequency, measured by the total number of stools passed during 24 and 48 hours from the initiation of treatment, and hospital duration, measured by the total duration of hospital stay in hours. The null hypothesis states that racecadotril combined with standard treatment has no effect on reducing the mean number of stools passed during 48 hours compared to standard treatment alone in pediatric patients with acute watery diarrhea, while the alternate hypothesis suggests that racecadotril combined with standard treatment will significantly reduce the mean number of stools passed during 48 hours compared to standard treatment alone in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized Patients with acute watery diarrhea of both genders who are

  1. Age: 03 months to 05 years
  2. Present in first 24 hours of onset of disease.

     Exclusion Criteria:

  <!-- -->

  1. Parenteral Diarrhea
  2. Chronic Diarrhea like Coeliac disease, Lactose intolerance
  3. Mal-absorption Syndromes
  4. Diarrhea related to food poisoning, dysentery as suggested by history
  5. Severe dehydration patents who are vitally unstable.
  6. Diarrhea associated with measles.
  7. Persistent vomiting
  8. Abdominal distention
  9. Patients allergic to racecadotril
  10. Patients managed before enrolled to study

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Estimated)
Dates: Start 2024-08-02 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
Stool frequency | 48 hours
  Total no. of stools passed during 24 and 48 hours from initiation of treatment will be compared between two groups

SECONDARY OUTCOMES:
Hospital Duration | 48 Hours
  Total duration of hospital stay taken in hours

IPD SHARING:
Plan to Share IPD: No